CLINICAL TRIAL: NCT01084512
Title: Phase 0 Study of Chest Wall Kinematics and Respiratory Muscle Action During Supine Breathing in Individuals With and Without Spinal Cord Injury.
Brief Title: Chest Wall Kinematics and Respiratory Muscle Action During Supine Breathing in Individuals With and Without Spinal Cord Injury
Acronym: SCI
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Kwan-Hwa Lin, National Taiwan University
Other Study IDs: 9461701293
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-02

CONDITIONS: Spinal Cord Injury
Keywords: kinematic analysis,; three-compartment model,; chest wall motion,; spinal cord injury.
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy group: control subjects
- Paraplegic group: Paraplegic subjects
- Tetraplegic group: tetraplegic subjects

SUMMARY:
Objective: To investigate the movement strategy of breathing based on three-compartment model measured by optoelectronic plethysmography (OEP) and electromyography (EMG ) among individuals with and without spinal cord injury in supine posture during deep inspiration.

Design: cross sectional repeated-measure with age matched control group. Setting: Motion Analysis Laboratory Participants: Seven tetraplegic and five paraplegic subjects and twelve age matched healthy controls were recruited.

Intervention: Not applicable.

DETAILED DESCRIPTION:
Main Outcome Measures: The volume changes of chest wall and respiratory electromyographic ( EMG ) muscle activity were measured simultaneously by OEP and surface EMG. The variables included volume changes (ΔV ), ratio of volume changes (ΔVr ), peak velocity of volume changes ( PV ), the percentage of peak velocity occurs ( PPV ) in three compartments (upper thorax, UT; lower thorax, LT; and abdominal compartment, AB), and Root Mean Square EMG ( RMS EMG ) of sternocleidomastoid and diaphragm (combined with intercostalmuscles).

Results: Ttetraplegic individuals had smallerΔVUT andΔVLT than those of control subjects(P< .006 and .006, respectively). Furthermore, the ΔVr of AB was greater than those of UT and LT( P< .006, .006, respectively), PVAB was smaller than PVLT ( P< .006), PPVUT was greater than PPVLT and PPVAB ( P< .008, .008, respectively ). The paraplegic subjects had smallerΔVLT than that of control subjects ( P< .006 ). ΔVr of UT was greater than that of LT, and both PVUT and PVAB were greater than PVLT ( P< .006 and .006, respectively). However, the paraplegic subjects preferred to all three compartments to achieve the maximal inspiration, like control group. In control group, onlyΔVAB was comparable with other compartments. ΔVr of UT was greater than LT, and PVUT was greater than PVLT and PVAB ( P<.006 and .006, respectively). For the RMS EMG, it demonstrated that average RMS EMG of two muscles in both tetraplegic and paraplegic group were greater than that in control group (P< .017 and .017, respectively).

Conclusion: The results applied the three-compartment model of chest wall to investigate the breathing pattern by OEP in individuals with and without SCI during inspiration of vital capacity breathing in supine posture. There were some interesting findings that (1) the tetraplegic subjects used AB contributed most volume changes, they can expand the AB more easily, and the UT took the responsibility to performed the final adjust during the inspiration; (2) the paraplegic subjects used UT contributed the most volume changes, they expanded the both UT and AB more easily, and all three compartment moved together during the inspiration; (3) the control subjects used UT to increase the most volume changes, they can expand UT more than the others, and all three compartments moved together during the inspiration phase, (4) the results of RMS EMG showed that the central neural drive in both tetraplegic and paraplegic subjects were greater than control group.

ELIGIBILITY:
Inclusion Criteria:

* (1) motor complete loss below level of injury with American Spinal Injury Association Classification (ASIA) class A or B19;
* (2) post-injury duration at least 0.5 year;
* (3) male subject due to high incidence rate in Taiwan20and the necessity of total exposure of the chest wall during the data collection.

Exclusion Criteria:

* (1) with any traumatic history of the chest wall,
* (2) with any respiratory disease and musculoskeletal problem that interfered with the experimental protocol;
* (3) having infections during the data collection period.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Chest wall motion | 6 months after spinal cord injury

SECONDARY OUTCOMES:
ultrasonography | 6 months after spinal cord injury

CONTACTS AND LOCATIONS:
Locations (1):
- School and graduate institute of physical therapy, Taipei, Taiwan, Taiwan